CLINICAL TRIAL: NCT00374829
Title: The Impact of a Multidisciplinary, Information Technology Supported Program on Blood Pressure Control in Primary Care (The Loyal Study)
Brief Title: Impact of an IT-Based and Healthcare Professional Support Program on Patients With High Blood Pressure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Université de Montréal (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRA 0530008; ISRCTN75436659
Record Dates: First submitted 2006-09-08; First posted 2006-09-12 (Estimated); Last update posted 2009-05-08 (Estimated); Status verified 2007-05

CONDITIONS: Hypertension
Keywords: randomised prospective trial; medication refill compliance; hypertension; ambulatory blood pressure monitoring; information technology based patient support system; process of care, quality of life, pharmacoeconomics; multidisciplinary patient management
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: An IT-based patient follow-up and reminder system

SUMMARY:
The study is a randomised controlled trial to evaluate the impact of a program using information technology (IT) and healthcare professional support in patients with high blood pressure (BP) compared to usual care. The program helps patients monitor their own BP and medication and keeps nurses,physicians and pharmacists informed while respecting patient confidentiality. The IT system links directly with the patient's pharmacy data. Using pharmacy data and responses to questions on compliance and BP control, the IT system provides appropriate counselling, telephone reminders, generates prescription refill and renewal reminder calls and monitors BP. The system reports compliance and self recorded BP measurements to healthcare providers and also links with a nurse. This is so that the nurse, the patient's doctor and pharmacist can help answer questions about medication and controlling high blood pressure.

A total of 500 patients in Laval, Quebec will participate in the study. Half of the patients will have the program plus usual care and the other have usual care only. We hypothesize that the program will improve BP control by helping patients take their medication properly and by helping doctors ensure that the best strength and kinds of medication are used to control high blood pressure. We believe the program will achieve this by helping to improve communication between patients and healthcare providers, without adversely impacting quality of life. Additional sub-studies will determine if the program is cost effective and can be applied in real practice and if the program helps patients, doctors, pharmacists and nurses communicate better.

DETAILED DESCRIPTION:
As the Canadian population ages, the number of hypertensive patients that have major cardiovascular events will increase, placing additional burden on healthcare resources. The positive effects of optimal blood pressure (BP) control on morbidity and mortality have been clearly established. In spite of this, data suggest that only 13% of Canadian hypertensive patients are adequately controlled. It is believed that much of this poor BP control can be attributed to: patient non-compliance; acceptance of inadequate BP control by clinicians; lower BP goals; and the fact that it is difficult to achieve adequate BP control with monotherapy in the majority of patients.

There is a recognised need to improve communication between patients and health care providers and among healthcare professionals themselves and to develop new tools to improve patients compliance. We have developed an information technology (IT)-based system to empower patients to be responsible for monitoring their blood pressure (BP) and compliance and to facilitate communication with healthcare providers. The IT-based system links with actual pharmacy prescription refill and renewal data. Using these data as well as responses to questions on compliance and BP control that patients provide using the telephone, the system: offers patients counselling and telephone reminders; generates prescription refill and renewal reminder calls; and, monitors patient recorded BP. The system generates monthly reports to the treating physician and pharmacist on compliance and blood pressure control, which we believe will help them monitor and modify therapy as appropriate. The system also links patients with a nurse if BP is inadequately controlled and/or if patients are non-compliant, who, in turn, can then provide appropriate counselling and refer the patients to their physician or pharmacist as appropriate.

The randomised controlled trial (RCT), is designed to determine if this multidisciplinary, information-technology supported hypertension management program (hereafter called "the intervention") will improve BP control. We hypothesise that the intervention will achieve this through enhanced compliance with pharmacotherapy by patients and the use of higher doses and more anti-hypertensive agents when appropriate, without adversely impacting quality of life. Additional sub-studies will be conducted to explore the perceptions patients, their families and healthcare providers have on the impact of the intervention on the process of care and to further explore the links between communication and relationship skills (CRS), compliance and health-care outcomes and to further evaluate collaborative models of inter-professional practice.

The primary outcome measure is to evaluate the impact of the intervention on the mean change in 24-hour systolic and diastolic BP levels measured using ABPM. Secondary objectives are to assess the likely mechanisms that account for the results for the primary objective by measuring: refill compliance to the BP lowering regimen, the number of dosage and/or type of medication changes over the 12-month study period and the time interval between prescriptions to initiate these changes, the number of different anti-hypertensive agents used and the number and nature of interventions by pharmacists, nurses and physicians. In addition average 24 hour and nocturnal diastolic and systolic blood pressure measurements using 24 hour continuous ABPM at 12-month follow-up; the proportion of subjects who achieve target BP according to the Canadian recommendations; the subject's health related quality of life at baseline and at 12-months; the cost-effectiveness of the system from a third party payer's perspective in terms of $ per QALY (derived from the EuroQoL) and $ per years of life gained, after modelling for long term reduction in events associated with better blood pressure control; the subject's acceptance or refusal of all or part of the IT-based reminder and blood pressure monitoring system; and, the physician's and subject's perception of the impact of the system on the process of care.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with untreated or suboptimally controlled hypertension
* Age equal to or greater than 18 years
* Ambulatory outpatients currently being treated in primary care setting
* Capable of giving informed consent
* Able to communicate in and read either French or English
* Purchase their medication at a pharmacy participating in the program
* Agree to stay with one pharmacy for the duration of the study
* Able to have a 24 hour ABPM recording within 7 days of screening
* Written informed consent obtained

Exclusion Criteria:

* Unlikely to complete study due to life-threatening disease or condition
* Having chronic atrial fibrillation
* Unable to use an ordinary telephone
* Pregnant at the initial visit
* Participating in another clinical trial concomitantly
* Participated in an antihypertensive clinical trial within the past 2 months
* Living with another subject that is currently participating in the study
* Delaying pharmacotherapy for baseline ABPM could put the subject at risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2004-05; Study Completion 2007-06 (Estimated)

PRIMARY OUTCOMES:
Change in the mean 24-hour systolic and diastolic BP using ABPM | 12 months

SECONDARY OUTCOMES:
Refill compliance to the BP lowering regimen | 12 months
Dosage and/or type of medication changes | 12 months
Change in the mean daytime and nocturnal systolic and diastolic BP between baseline and 12 months measured using ABPM | 12 months
Proportion of subjects who achieve target BP | 12 months
Proportion of patients presenting with an adverse cardiovascular event | 12 months
The mean change in health related quality of life | 12 months
Number and nature of pharmacist, nurse and physician interventions | 12 months
Long-term cost-effectiveness of the system | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Rinfret, MD MSc FRCPC, Principal Investigator — Centre de Recherche, Centre Hospitalier de l'Université de Montréal (CRCHUM); Pavel Hamet, MD PhD FRCPC, Study Director — Centre de Recherche, Centre Hospitalier de l'Université de Montréal (CRCHUM)
Locations (1):
- Cité de la Santé de Laval, Laval, Quebec, Canada

REFERENCES:
- [Derived] Rinfret S, Lussier MT, Peirce A, Duhamel F, Cossette S, Lalonde L, Tremblay C, Guertin MC, LeLorier J, Turgeon J, Hamet P; LOYAL Study Investigators. The impact of a multidisciplinary information technology-supported program on blood pressure control in primary care. Circ Cardiovasc Qual Outcomes. 2009 May;2(3):170-7. doi: 10.1161/CIRCOUTCOMES.108.823765. Epub 2009 May 5. PMID 20031834
- See also: ISRCTN Register — http://www.controlled-trials.com/